CLINICAL TRIAL: NCT05064137
Title: Clinical Efficacy of Different Remineralizing Agents in Treatment of White Spot Lesions Among a Group of Egyptian Children : A Randomized Clinical Trial
Brief Title: Clinical Efficacy of Different Remineralizing Agents in Treatment of White Spot Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yara Ahmed Ibrahim Abdellatif, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 257
Record Dates: First submitted 2021-09-18; First posted 2021-10-01 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Remineralization
MeSH Terms: interventions — Sodium Fluoride

STUDY DESIGN:
Who Masked: Participant
Masking Description: Double blinded ( participant and statistician )
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Curodont Repair® ( monomeric self - assembling peptide P11-4 ) (Experimental): Self assembling peptide P11-4 as Curodont Repair® can remineralize WSLs in a deeper manner than fluoride by guided enamel regeneration by forming a three-dimensional matrix within the subsurface body of an initial carious lesion to which calcium and phosphate ions found in natural saliva can bind and build de novo hydroxyapatite crystals.
  Interventions: Drug: Monomeric self - assembling peptide P11-4
- Clinpro white varnish® ( Tricalcium Phosphate Fluoride Varnish, 5% F- ) (Experimental): Tri-calcium phosphate can be hydrolyzed rapidly to form calcium hydroxyapatite (HAp). The processes of hydrolysis and formation of HAp are accelerated by the presence of NaF ions as in case of Clinpro white varnish®. Moreover, the HAp formed by such hydrolysis tends to have a greater uptake of fluoride than conventional HAp.
  Interventions: Drug: Tricalcium phosphate fluoride varnish, 5% F-
- Voco-profluorid® fluoride varnish (5% sodium fluoride) (Active Comparator): Fluoride varnish is the gold standard for treating WSLs.
  Interventions: Drug: fluoride varnish (5% sodium fluoride)

INTERVENTIONS:
Drug: Monomeric self - assembling peptide P11-4 — Monomeric self - assembling peptide P11-4 ( Curodont Repair ) is a remineralizing agent applied on tooth surface after treating it with 3% sodium hypochlorite for 20 seconds then etching it with 37% phosphoric acid for 20 seconds followed by rinsing then dryness.
  Other Names: Curodont Repair
  Arms: Curodont Repair® ( monomeric self - assembling peptide P11-4 )
Drug: Tricalcium phosphate fluoride varnish, 5% F- — Tricalcium phosphate fluoride varnish, 5% F- ( Clinpro White Varnish ) is a remineralizing agent applied on tooth surface after mixing it with a brush onto the dosage guide.
  Other Names: 3M Clinpro white varnish
  Arms: Clinpro white varnish® ( Tricalcium Phosphate Fluoride Varnish, 5% F- )
Drug: fluoride varnish (5% sodium fluoride) — fluoride varnish (5% sodium fluoride) ( Voco-profluorid ) is a remineralizing agent applied on tooth surface then area is allowed to become wet (either by gentle rinsing or natural salivary flow) to ensure setting of VOCO Profluorid Varnish.
  Other Names: Voco-profluorid
  Arms: Voco-profluorid® fluoride varnish (5% sodium fluoride)

SUMMARY:
The aim of the present study is to evaluate the efficiency of Self-assembling Peptide P11-4, Tricalcium Phosphate Fluoride Varnish, 5% F- and 5% fluoride varnish in remineralization of WSLs in primary dentition among a group of Egyptian children.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy cooperative children
* Aging from 3-5 years old child
* Both genders
* Primary teeth with active WSLs on buccal or labial surfaces
* Patient and parent acceptance to treatment and maintenance of good oral hygiene

Exclusion Criteria:

* Restored teeth
* White spot lesions due to fluorosis
* Teeth with hypoplasia
* Lesions that require an invasive treatment
* Any pathology or concomitant medication affecting salivary flow or causing dry mouth

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Size of WSL ( white spot lesion ) | through study completion, an average of 8 months
  Size of WSL measured by scored dental probe

SECONDARY OUTCOMES:
Regression of caries | through study completion, an average of 8 months
  Regression of caries evaluated by International Caries Detection and Assessment System (ICDAS) II
Inactivation of active carious lesions | through study completion, an average of 8 months
  Inactivation of active carious lesions evaluated by Lesion activity assessment (LAA-ICDAS)
Mineral content of WSL | through study completion, an average of 8 months
  Mineral content of WSL measured by fluorescence camera VistaCam iX